CLINICAL TRIAL: NCT02622373
Title: Impact of Currently Recommended Postnatal Nutrition on Neonatal Body Composition
Status: Completed | Type: Observational
Sponsor: Vishal Pandey, M.D. (Other)
Responsible Party: Sponsor-Investigator, Vishal Pandey, M.D., Assistant Professor, Department of Pediatrics, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: STUDY00002323
Record Dates: First submitted 2015-11-16; First posted 2015-12-04 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Premature Birth; Preterm Birth
Keywords: Pea Pod; Body composition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Birth Between 23-32 Weeks Gestation: Babies born between 23-32 weeks of gestational age will have their body composition determined using PEA POD Infant Body Composition System at 34 weeks, 36 weeks and 40 weeks of corrected age.
  Interventions: Device: PEA POD Infant Body Composition System
- Birth Between 34-36 Weeks Gestation: Babies born at 34 weeks and 36 weeks of gestational age will have their body composition measured using PEA POD Infant Body Composition System as soon as they are off parenteral nutrition and receiving full enteral nutrition.
  Interventions: Device: PEA POD Infant Body Composition System
- Birth at Term: Body composition will be measured using PEA POD Infant Body Composition System in this group will be obtained prior to discharge.
  Interventions: Device: PEA POD Infant Body Composition System

INTERVENTIONS:
Device: PEA POD Infant Body Composition System — The non-invasive device used in this study to measure a baby's body composition is a called a Pea Pod. The Pea Pod is a quick, safe, non-invasive and reliable bedside procedure used to measure changes in infant body composition.

SUMMARY:
The purpose of this study is to gain information that may be useful in helping to figure out better or newer ways to provide nutrition to babies born premature.

DETAILED DESCRIPTION:
Babies born premature weigh significantly less at the time of hospital discharge when compared to babies born at the corresponding age. The researchers in this study believe that the lower body weight at discharge may be due to lower muscle mass. However, there is no such information available for that at this time. It is important to have this information as babies who weigh less than normal at hospital discharge may develop higher blood pressure and higher sugar levels when they are 10-15 years old.

By doing this study, researchers will be able to have information about the baby's muscle mass, which will help the researchers to provide better nutrition to babies who are born premature. Researchers will also be able to determine if there are any differences in the muscle/fat mass based on the type of feeding (breast milk alone, formula alone or a combination of breast milk and formula). This information may be beneficial in helping to promote the appropriate type of feeding for babies born premature.

ELIGIBILITY:
Inclusion Criteria:

* Newborns <32 weeks gestational age, singleton or multiple gestation
* 34-36 weeks gestational age newborns
* Term healthy infants from uncomplicated pregnancy

Exclusion Criteria:

* Babies with life threatening illness unlikely to survive
* Congenital and chromosomal anomalies

Ages: 23 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study group involves premature infants born between 23 to 32 weeks gestation, while babies born at 34 weeks, 36 weeks and ≥37 and ≤ 42 weeks gestational age will serve as control groups.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in the Fat mass percentage between 36 and 40 weeks in preterm infants | Change in the Fat mass percentage between 36 weeks and 40 weeks corrected age
  Body composition as determined by the PEA POD air displacement plathesmography would determine the fat mass percentage and the serial measure of this parameter would determine the changes in the fat mass percentage indicating the quality of growth between 36 and 40 weeks post conceptional age. At 40 weeks corrected age, the fat mass percentage of the premature infants would be compared with ten healthy term infants born to healthy mothers with uncomplicated pregnancies.

SECONDARY OUTCOMES:
Comparison of the Fat mass percent between preterm infants at 40 weeks and those born at Term gestation. | 40 weeks corrected age
  The Fat mass percentage in preterm infants at the 40 weeks corrected age would be compared with healthy full term infants born following an uncomplicated pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Pandey, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Simon L, Frondas-Chauty A, Senterre T, Flamant C, Darmaun D, Roze JC. Determinants of body composition in preterm infants at the time of hospital discharge. Am J Clin Nutr. 2014 Jul;100(1):98-104. doi: 10.3945/ajcn.113.080945. Epub 2014 May 7. PMID 24808483